CLINICAL TRIAL: NCT05241015
Title: Investigation of the Effect of Sensorimotor Training on Upper Extremity Functions, Activity and Participation in Parkinson's Patients
Brief Title: Effect of Sensorimotor Training on Upper Extremity in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: TC Erciyes University (Other); Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Ozlem Menevse, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/295 (Erciyes University)
Record Dates: First submitted 2022-01-07; First posted 2022-02-15 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Upper Extremity; Sensorimotor Training; ICF; Function
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive standard physiotherapy program used for PD will be applied, 3 times a week for 8 weeks.
  Interventions: Other: Control Group
- Exercises Group (Experimental): In addition to standard physiotherapy programme, patients in this group will also receive sensorimotor training.
  Interventions: Other: Exercises Group

INTERVENTIONS:
Other: Control Group — Treatment protocol; It will be applied to improve posture, strengthen muscles, eliminate shortness, increase flexibility, balance/coordination, sit up/stand up and in-bed mobilization, and improve gait. Before taking the treatment, a general evaluation will be made and as a result of this evaluation, muscle shortness, loss of strength, postural disorders and the activities and positions they have the most difficulty in daily life will be determined. Treatment programs will be shaped according to the problems determined in line with the evaluations made.
  Arms: Control Group
Other: Exercises Group — In addition to the standard physiotherapy program, sensorimotor training including the cervical region will be given to the this group. Deep cervical flexor and extensor muscles, which provide stability in the cervical region, will be trained. A Pressure Biofeedback Device will be used to train the deep cervical flexors. Both positional and kinesthetic sensory training will be provided by maintaining the stability of the cervical region by means of the laser kit that provides visual feedback.Additionally, oculomotor exercises will be given.
  Arms: Exercises Group

SUMMARY:
There are many factors affecting the upper extremity such as tremor, bradykinesia, rigidity, and postural instability in Parkinson's patients. According to the International Classification of Functioning, Disability and Health (ICF) model, there are restrictions on people's activities and participation in life due to structural and functional disorders affecting the upper extremity in PD.

In PD, integrating and using proprioceptive feedback, sensorimotor integration and peripheral sensory functions are reported to be impaired. Numerous studies show that the main source of motor problems in PD is dysfunction of sensorimotor integration. Since the cervical region contains a dense concentration of proprioceptive organs such as muscle spindles, it plays an important role in providing afferent proprioceptive information for postural control. Therefore, sensorimotor training targeting the cervical region gains importance. In this study, we aim to reduce PD-specific upper extremity disorders and related activity and participation limitations by increasing motor control in the cervical region with sensorimotor training. Patients with Parkinson's disease will be included in the study and randomly divided into 2 groups. While the general physiotherapy program will be applied to the control group, sensorimotor training will be given in addition to the exercise group.

ELIGIBILITY:
Inclusion Criteria:

* Having idiopathic Parkinson's disease over the age of 40
* Meets the diagnostic criteria of the United Kingdom Parkinson's Disease Society Brain Bank
* Hoehn-Yahr Staging <3
* Mini mental test score of 24 and above
* In the "on" period
* Receiving oral therapy only

Exclusion Criteria:

* Patients receiving device-assisted therapy
* Patients receiving apomorphine therapy
* Patients with mini mental test scores below 24
* Patients who use drugs (antidepressants, etc.) that will affect cognitive functions
* Patients with hearing and speech problems
* Patients with orthopedic, neurological and vestibular problems other than Parkinson's that may prevent them from completing the tests and treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Posture Analysis | Change from baseline at 8 week
  New York Posture Rating Chart
Tremor | Change from baseline at 8 week
  Fahn; Tolosa, Marin Clinical Tremor Rating Scale will be used to evaluate tremor. Each item was scored between 0-4. A lower score is an indicator of better status.
Unified Parkinson's Disease Rating Scale | Change from baseline at 8 week
  Unified Parkinson's Disease Rating Scale is a scale that evaluates disability and disorders related to Parkinson's and consists of 4 main subtitles and 42 questions in total . Each item was scored between 0-4 . A lower score is an indicator of better status.
Proprioception | Change from baseline at 8 week
  For proprioception, joint position error in the cervical region and upper extremity will be evaluated with the laser kit.
Tactile acuity | Change from baseline at 8 week
  For upper extremity tactile acuity, moving 2-point discrimination test (MTPD) will be performed using an esthesiometer.
Touch threshold | Change from baseline at 8 week
  Semmes Weinstein Monofilament Test will be used to evaluate upper extremity touch threshold.
Pain threshold | Change from baseline at 8 week
  Algometer will be used to evaluate upper extremity pain threshold.
Pain intensity | Change from baseline at 8 week
  Visual pain scale (VAS) will be used to evaluate upper extremity pain.In the evaluation, pain averages ranging from 0 to 10 cm are given. "0" indicates that there is no pain, while as the score increases, the severity of pain increases.
Hand Grip Strength | Change from baseline at 8 week
  Hand Dynamometer will be used to measure hand grip strength.
Pinch Grip Strength | Change from baseline at 8 week
  Pinch meter will be used to measure pinch grip strength.
Endurance of Cervical Muscles | Change from baseline at 8 week
  Craniocervical Flexion (CSF) test, Evaluation of cervical flexor-extensor muscles
Fatigue | Change from baseline at 8 week
  Parkinson's Fatigue Scale will be used to evaluate fatigue. It is consists of 16 items related to presence of fatigue. All items are scored by patients using a five-point Likert-type scale including response options ranging from '(1) strongly disagree' to '(5) strongly agree'. A higher score indicates a higher level of fatigue.
Hand functions | Change from baseline at 8 week
  Purdue Pegboard Test (PPT)
Dual Task Performance | Change from baseline at 8 week
  During the Purdue Pegboard Test, the second task will be added and the completion time will be recorded.
Disabilities of the Arm, Shoulder and Hand Questionnaire | Change from baseline at 8 week
  It will be used to determine the problems experienced in the use of the upper extremity. It consists of 3 sections. All questions are answered according to a 5-point Likert system. A score between 0-100 is obtained from each section. The higher the score, the higher the disability.
Quality of life evaluation | Change from baseline at 8 week
  Parkinson's Disease Questionnaire (PDQ-39) will be used to evaluate quality of life. It contains 39 items in total. A score between 0 and 4 is given for each question. A high overall score indicates worsening quality of life.
Evaluation of Environmental Factors | Change from baseline at 8 week
  Questions structured by the researchers will be used on the issues of support and attitudes under the environmental factors heading of the ICF model. Questions are scored between 0 and 10. A high score indicates high satisfaction.
Motor speed | Change from baseline at 8 week
  Motor speed will be evaluated using the Finger tapping test.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Department of Physiotherapy and Rehabilitation, Kayseri, Turkey (Türkiye)